CLINICAL TRIAL: NCT05314660
Title: Arresting Active Dentine Lesions and Quality of Life Among a Group of Preschool Children in Mansoura City.
Brief Title: Arresting Active Dentine Lesions and Quality of Life Among a Group of Preschool Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A22080120
Record Dates: First submitted 2022-03-24; First posted 2022-04-06 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2020-01

CONDITIONS: Caries Arrest
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: 3 equal groups receiving 3 different protocols
Masking Description: The operator must know the group in which the participant is enrolled so as to provide and carry out the intended treatment protocol. Randomization was preformed by block randomization by the nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Silver diamine fluoride group (Experimental): Application of 38% SDF.
  Interventions: Drug: 38 % silver diamine fluoride
- Atrumatic restorative technique (Experimental)
  Interventions: Procedure: Atraumatic restorative technique
- Ultra conservative treatment (UCT) (Experimental)
  Interventions: Procedure: Ultra conservative dentistry

INTERVENTIONS:
Drug: 38 % silver diamine fluoride — Application of 38% SDF on carious dentine lesions.
  Arms: Silver diamine fluoride group
Procedure: Atraumatic restorative technique — Hand excavation of carious dentine followed by application of Glass ionomer
  Arms: Atrumatic restorative technique
Procedure: Ultra conservative dentistry — Removal of soft dentine and enlarging of cavity to control bio film
  Arms: Ultra conservative treatment (UCT)

SUMMARY:
Testing 3 different caries arresting techniques and the quality of life of a group of preschool children in Mansoura city, Egypt.

DETAILED DESCRIPTION:
135 preschoolers were allocated randomly into 3 groups to receive 3 techniques to evaluate caries arrestment. The first group received 38% silver diamine fluoride, the second received conventional Atraumatic restorative technique and the third group received ultra consevative treatment (UCT). The subjects were followed up at 3, 6 and 12 months to check caries activity according to the ICDAS.

The parents of the children answered the Arabic ECOHIS before treatment and after 3 months to assess oral health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* healthy children aged 3-5
* residents of mansoura city
* having at least one carious dentine lesion

Exclusion Criteria:

* large carious lesions approximating the pulp
* signs of pulpitis, fistula, abscess.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Caries arrestment assessed by the International caries detection and assessment system (ICDAS) and absence of pain and signs of pulpal involvement. | 1 year
  Absence of pains and signs of pulpal involvement and caries classified as inactive by ICDAS was considered a successful outcome. When the lesions appeared shiny and felt hard on probing (for SDF and UCT). For ART success was measures by the presence of intact restoration and avsence of pain.

SECONDARY OUTCOMES:
Early childhood oral health impact scale (ECOHIS) | 3 months
  Comprises 13 questions of four domains; child symptoms, function, pscychology and social interactions. Questionnaire answered at the first appointment and 21 days later. Lowest score is 0, highest is 52 and higher score indicates poor oral health related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Basma Hamza, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data regarding the A-ECOHIS will be available to share if needed

REFERENCES:
- [Derived] Hamza BE, Attia NM, Abdellatif AM, Hegazy SA. Arresting Active Carious Lesions Using Minimal Intervention Dentistry among a Group of Preschool Children: A Randomized Controlled Clinical Trial. Int J Clin Pediatr Dent. 2024 Sep;17(9):1018-1024. doi: 10.5005/jp-journals-10005-2927. PMID 39664835